CLINICAL TRIAL: NCT00411632
Title: A Phase II Study of Erlotinib (Tarceva) in Combination With Bexarotene (Targretin) in Chemorefractory Patients With Advanced Non-Small Cell Lung Cancer (NSCLC)
Brief Title: BATTLE Program: Tarceva and Targretin in Patients With Advanced Non-Small Cell Lung Cancer (NSCLC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2005-0826; NCI-2012-02089 (Registry Identifier: NCI CTRP); W81XWH-06-1-0303 (Other: Department of Defense)
Record Dates: First submitted 2006-12-12; First posted 2006-12-14 (Estimated); Results first posted 2020-01-21 (Actual); Last update posted 2020-01-29 (Actual); Status verified 2020-01

CONDITIONS: Lung Cancer
Keywords: Lung Cancer; Non-Small Cell Lung Cancer; NSCLC; Erlotinib; Tarceva; Bexarotene; Targretin; OSI-774; Battle Program
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Bexarotene; Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Bexarotene + Erlotinib (Experimental): Bexarotene 400 mg/m^2 by mouth daily x 28 Days. Erlotinib 150 mg by mouth daily x 28 Days.
  Interventions: Drug: Bexarotene; Drug: Erlotinib

INTERVENTIONS:
Drug: Bexarotene — 400 mg/m^2 by mouth daily x 28 Days
  Other Names: Targretin
Drug: Erlotinib — 150 mg by mouth daily x 28 Days
  Other Names: Tarceva; OSI-774

SUMMARY:
The goal of this clinical research study is to evaluate the effectiveness of Tarceva® (OSI-774, erlotinib hydrochloride) in combination with Targretin® (bexarotene) in treating NSCLC. The safety of this treatment will also be studied, as well as the treatment's effect on different cells in the body and the participants' overall response.

DETAILED DESCRIPTION:
Erlotinib hydrochloride is designed to help block the activity of an enzyme that is believed to play an important role in cell growth. Researchers want to find out if blocking these enzymes will slow tumor growth. Bexarotene is designed to control cancer cell growth and division.

In order to enroll in this study, you must also be enrolled in Protocol 2005-0823 (NCT00409968): A Biomarker-integrated study in Chemorefractory Patients with Advanced Non-Small Cell Lung Cancer. Protocol 2005-0823 (NCT00409968) is the screening study in a group of studies called the BATTLE program. Participants in Protocol 2005-0823(NCT00409968) are assigned to one of the research studies. The results of your tumor analysis helped the study doctor determine to assign you to this particular research study.

While on study, you will take erlotinib hydrochloride and bexarotene by mouth once a day. Erlotinib hydrochloride tablets should be taken preferably in the morning 1 hour before or 2 hours after a meal with no more than 7 ounces of water. If you forget to take a dose, the last missed dose should be taken as soon as you remember, as long as it is at least 12 hours before the next dose is due to be taken. The next day, you should take the scheduled dose at the usual time.

Bexarotene capsules should be taken with or immediately after a meal. If you miss a dose, take it as soon as possible, with food. However, if it is nearly time for your next dose, skip the missed dose and continue your dose schedule as before.

Every attempt should be made to keep from vomiting the medication for at least 30 minutes after taking it. For example, if you feel nauseated before or after taking the medication, anti-nausea medications should be used.

The erlotinib hydrochloride tablets and bexarotene capsules should be stored at room temperature. Bexarotene capsules should not be stored near heating devices, high temperatures or humidity, or where children or pets have access to them. Bexarotene capsules should be protected from sunlight.

Every 4 weeks (1 cycle) your medical history will be recorded and you will have a physical exam, including measurement of vital signs (blood pressure, pulse, temperature, and breathing rate) and weight. You will have routine blood tests (about 2 teaspoons) and a performance status evaluation (questions about your ability to perform everyday activities). You will have blood drawn (about 1-2 teaspoons) to check you thyroid function. You will also have blood drawn (about 1-2 teaspoons) to check your lipid profile weekly for the first 4 weeks and then every cycle after that. Your study doctor will also ask you about any medications you are taking and your smoking history.

Every 2 cycles, your tumor will be evaluated by chest x-ray and computed tomography (CT) or magnetic resonance imaging (MRI) scans to evaluate the status of the disease. If you are taking Coumadin® (warfarin), you will have blood drawn (about 1-2 teaspoons) to check your blood clotting function weekly for the first 5 weeks of treatment and then every cycle after that.

You may continue receiving erlotinib hydrochloride and bexarotene for as long as the cancer responds to study treatment. Your doctor may decide to take you off this study if you experience intolerable side effects, your medical condition gets worse, or you are unable to comply with study requirements. If you stop study treatment, you may be able to enroll in 1 of the remaining 3 protocols of the BATTLE program.

After you have stopped taking the study treatment, you will have a physical exam, including measurement of vital signs. Blood (about 2 teaspoons) and urine will be collected for routine tests. You will also have blood drawn (about 1-2 teaspoons) to check your blood clotting function. You will have a performance status evaluation, a chest x-ray, and a CT or MRI scan. Following this evaluation, you will be contacted by telephone every 3 months for up to 3 years, to see how you are doing.

This is an investigational study. Erlotinib hydrochloride is approved by the FDA for treatment of NSCLC in patients who have relapsed. Bexarotene is approved by the FDA for the treatment of cutaneous T-cell lymphoma (CTCL). Their use together in this study is investigational. Up to 72 patients will take part in this multicenter study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. The patient has a diagnosis of pathologically confirmed NSCLC by tumor biopsy and/or fine-needle aspiration.
2. The patient has a diagnosis of either stage IIIB, stage IV, or advanced, incurable NSCLC, and failed at least one front-line metastatic NSCLC chemotherapy regimen. (Patients who have failed adjuvant or locally advanced therapy within 6 months are also eligible to participate in study).
3. The patient has uni-dimensionally measurable NSCLC.
4. Karnofsky performance status >/= 60 or ECOG performance status 0-2
5. The patient has biopsy accessible tumor.
6. The patient has adequate hematologic function as defined by an absolute neutrophil count (ANC) >/= 1,500/mm^3, platelet count >/= 100,000/mm^3, WBC >/= 3,000/ mm^3, and hemoglobin >/= 9 g/dL.
7. The patient has adequate hepatic function as defined by a total bilirubin level </= 1.5 X the upper limit of normal, and alkaline phosphatase, AST or ALT </= 2.5 X the upper limit of normal.
8. The patient has adequate renal function as defined by a serum creatinine level </= 1.5 mg/dL or a calculated creatinine clearance of >/= 60cc/minute.
9. The patient has PT < 1.5 x upper limit of normal
10. If patient has brain metastasis, they must have been stable (treated or asymptomatic) for at least 4 weeks after radiation if treated with radiation and not have used steroids for at least 1 week.
11. The patient is >/= 18 years of age.
12. The patient has signed informed consent.
13. The patient is eligible if disease free from a previously treated malignancy, other than a previous NSCLC, for greater than two years. Patients with a history of prior basal cell carcinoma of the skin or pre-invasive carcinoma of the cervix are exempt from exclusion.
14. Women of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Childbearing potential will be defined as women who have had menses within the past 12 months, who have not had tubal ligation or bilateral oophorectomy. Should a woman become pregnant or suspect that she is pregnant while participating in this study, she should inform her treating physician immediately. The patient, if a man, agrees to use effective contraception or abstinence.
15. Subject must be considered legally capable of providing his or her own consent for participation in this study.

Exclusion Criteria:

1. The patient has received prior investigational therapy, chemotherapy, surgery, or radiotherapy within 4 weeks of initiating study drug
2. The patient has undergone prior thoracic or abdominal surgery within 28 days of study entry, excluding prior diagnostic biopsy.
3. The patient has received radiation therapy to the measurable tumor within 6 months. Patients are allowed to have local irradiation for the management of tumor-related symptoms (bones, brain). However, if a patient has active new disease growing in the previously irradiated site, the patient will be eligible to participate in the study.
4. The patient has a significant medical history or unstable medical condition (unstable systemic disease: congestive heart failure (New York Heart Association Functional Classification class II or worse), recent myocardial infarction within 3 months, unstable angina, active infection (i.e. currently treated with antibiotics), uncontrolled hypertension). Patients with controlled diabetes will be allowed. Patient must be able to undergo procedure for tissue acquisition.
5. The patient has uncontrolled seizure disorder, active neurologic disease, or neuropathy >/= grade 2. Patients with meningeal or CNS involvement by tumor are eligible for the study if the above exclusion criteria are not met.
6. The patient is pregnant (confirmed by serum b-HCG if applicable) or is breastfeeding.
7. The patient has a concurrent condition which in the investigator's opinion makes it undesirable for the patient to participate in the trial or which would jeopardize compliance with the protocol.
8. The patient is actively taking herbal remedies or over-the-counter biologics (e.g., shark cartilage, high dose antioxidants).
9. Patients will be allowed to have prior biologic (i.e. VEGF, EGFR, etc.) therapy. However, the patient will be excluded from a given study if he/she has received the same therapy as the clinical trial (i.e. If a patient has been previously treated with bevacizumab, they are allowed to enroll in any of the 4 studies. If a patient has been previously treated with erlotinib, they are excluded from the clinical trials with erlotinib). In addition, if a patient has been previously treated with gefitinib (Iressa), they are excluded from the clinical trials with erlotinib.
10. The patient has dysphagia and who is unable to swallow intact capsules.
11. The patient has active gastrointestinal disease or a disorder that alters gastrointestinal motility or absorption (i.e., lack of integrity of the gastrointestinal tract such as a significant surgical resection of the stomach or small bowel).
12. The patient has received prior retinoid derivative therapy.
13. The patient has triglycerides >200.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2006-11-29 (Actual); Primary Completion 2018-02-23 (Actual); Study Completion 2018-02-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vali Papadimitrakopoulou, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Tam AL, Kim ES, Lee JJ, Ensor JE, Hicks ME, Tang X, Blumenschein GR, Alden CM, Erasmus JJ, Tsao A, Lippman SM, Hong WK, Wistuba II, Gupta S. Feasibility of image-guided transthoracic core-needle biopsy in the BATTLE lung trial. J Thorac Oncol. 2013 Apr;8(4):436-42. doi: 10.1097/JTO.0b013e318287c91e. PMID 23442309
- [Derived] Kim ES, Herbst RS, Wistuba II, Lee JJ, Blumenschein GR Jr, Tsao A, Stewart DJ, Hicks ME, Erasmus J Jr, Gupta S, Alden CM, Liu S, Tang X, Khuri FR, Tran HT, Johnson BE, Heymach JV, Mao L, Fossella F, Kies MS, Papadimitrakopoulou V, Davis SE, Lippman SM, Hong WK. The BATTLE trial: personalizing therapy for lung cancer. Cancer Discov. 2011 Jun;1(1):44-53. doi: 10.1158/2159-8274.CD-10-0010. Epub 2011 Jun 1. PMID 22586319
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Thirty-seven (37) patients were registered into this trial. All thirty-seven (37) patients were eligible to participate in this trial.
Pre-assignment Details: Participants enrolling in this study must first be enrolled in the BATTLE umbrella protocol and must meet all of the BATTLE eligibility criteria. Participants enrolled in the BATTLE program will be assigned to a specific biomarker-integrated study based on the adaptive randomization model.
Groups:
- Erlotinib + Bexatrtene: Bexarotene 400 mg/m^2 by mouth daily x 28 Days. Erlotinib 150 mg by mouth daily x 28 Days.
  Bexarotene: 400 mg/m^2 by mouth daily x 28 Days
  Erlotinib: 150 mg by mouth daily x 28 Days
Period: Overall Study
Arm/Group | Erlotinib + Bexatrtene
Started | 37
Completed | 36
Not Completed | 1
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Arm/Group | Bexarotene + Erlotinib
Number analyzed (Participants) | 37
Age, Continuous [Mean (Full Range); unit: years] | 62 [26 to 84]
Age, Customized [Count of Participants; unit: Participants]
  <=50 years | 6
  51-60 years | 11
  61-70 years | 11
  >70 years | 9
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 25
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 31
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 37

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With 8-week Progression-Free Survival (i.e. Disease Control Rate) Stratified by Cancer Mutation Type
Description: The primary objective is to determine the 8 week progression-free survival rate (i.e. disease control rate) in patients with advanced NSCLC who have failed at least one prior chemotherapy regimen. A radiologist independently assessed DC, which was defined as a complete or partial response or stable disease according to the RECIST(29) at the end of 8 weeks (start of treatment to end of second treatment cycle). PFS was assessed from the date of randomization to the earliest sign of disease progression or death from any cause. OS was assessed from the date of randomization until death from any cause. Tumor response was assessed every 8 weeks until disease progression. Toxicity was assessed in accordance with the National Cancer Institute Common Terminology Criteria for Adverse Events, version 3.0.
Time Frame: 8 weeks
Population: The primary end point was the 8-week DCR [complete or partial response or stable disease via Response Evaluation Criteria in Solid Tumors (RECIST, which we compared with the historical 30% DCR estimate in similar patients. Treatment efficacy (a positive finding) was defined as >0.80 probability of achieving>30% DCR.
Measure: Number; unit: participants
Groups:
- Erlotinib + Bexatrtene: Erlotinib 150 mg by mouth daily + bexarotene 400 mg/m2/day daily (1 cycle =4 weeks) for 2 cycles, tumor response will be evaluated at the end of the second cycle. Patients who have progressed stop treatment and can renter the main BATTLE protocol and be assigned to another Phase II trial.
Arm/Group | Erlotinib + Bexatrtene
Number analyzed (Participants) | 37
participants
  EGFR | 11
  KRAS/BRAF | 1
  VEGF/VEGFR-2 | 0
  RXR/Cyclin D1 | 1
  None | 5

ADVERSE EVENTS:
Time Frame: January 1, 2007 to November 24, 2009 Participants were assessed for response until progression and for survival up to 3 years following completion of study treatment.
Arm/Group | Erlotinib + Bexatrtene
All-Cause Mortality (participants affected / at risk) | 1/37
Serious Adverse Events (participants affected / at risk) | 8/37
Other Adverse Events (participants affected / at risk) | 13/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Erlotinib + Bexatrtene (N=37)
Hypertriglyceridema (Metabolism and nutrition disorders) | 4
Lipase increased (Investigations) | 1
Fatigue (Investigations) | 6
INR (Investigations) | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Erlotinib + Bexatrtene (N=37)
Hypertriglceridemia (Metabolism and nutrition disorders) | 8
Acne (Skin and subcutaneous tissue disorders) | 2
Hypothyroidism (Endocrine disorders) | 3
Diarrhea (Gastrointestinal disorders) | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-07-10): https://cdn.clinicaltrials.gov/large-docs/32/NCT00411632/Prot_SAP_000.pdf